CLINICAL TRIAL: NCT03990805
Title: Multi-center, Randomized, Double-Blind, Placebo Controlled Phase 3 Clinical Trial to Evaluate Efficacy and Safty of Mesenchymal Stem Cells JointStem in Patients With Knee Osteoarthritis
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of JointStem in Treatment of Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSR-CTph3-JS1
Record Dates: First submitted 2019-06-13; First posted 2019-06-19 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Degenerative Arthritis; Knee Osteoarthritis
Keywords: Stem Cell; Adipose tissue derived mesenchymal stem cell; osteoarthritis; degenerative arthritis; biostar; Rbio
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JOINTSTEM (Experimental): Autologous Adipose Tissue derived MSCs
  Interventions: Biological: JOINTSTEM
- saline (Placebo Comparator): saline
  Interventions: Drug: saline

INTERVENTIONS:
Biological: JOINTSTEM — JOINTSTEM Autologous Adipose Tissue derived MSCs 1x10^8cells/(saline), 1 time injection
  Other Names: Autologous Adipose Tissue derived MSCs
  Arms: JOINTSTEM
Drug: saline — saline, 1 time injection
  Arms: saline

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of autologous Adipose Tissue derived Mesenchymal stem cells (JOINTSTEM®) in patient with severe Knee Osteoarthritis.

DETAILED DESCRIPTION:
JOINTSTEM is injectables for an OA treatment that uses autologous adipose-derived mesenchymal stem cells. As it does not use allogenic tissues and is cultured without additional genetic modification, it is classified as 'autologous cell therapy' and is completely free of immunologic rejection.

It primarily aims to improve joint function. The intra-articular injection of JOINTSTEM is expected to stimulate the regeneration of cartilage, and to innovatively improve joint function with cartilage regeneration.

The subjects of this therapy were patients with K&L grade 3 aged 20 or older.

This study is a double-blind, randomized, placebo controlled study with two arms to evaluate JOINTSTEM as a treatment for subjects with osteoarthritis. Following a 2-week screening period, approximately 260 patients will be randomly assigned into one of the following two arms in a 1:1 ratio (1 JointStem : 1 placebo control). After each patient completes 6-month visit (Visit 5) and the data management team confirms all data have no issue, the individual database will be locked and the blinding will be open for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 and older, male and female
2. Patients must consent in writing to participate in the study by signing and dating an informed consent document
3. Diagnosis of degenerative arthritis of class 1-3 by ACR(American College of Rheumatology Criteria) Global functional criteria
4. Diagnosis of Kellgren and Lawrence grade 3 by radiographic criteria
5. Patients suitable for one of three conditions of 'diagnostic criteria for osteoarthritis of knee' based on ACR guideline

   * clinical and inspectional opinion
   * clinical and radiographic opinion
   * clinical opinion
6. Patients who has joint pain ≥ 50mm on 100mm VAS (Visual Analog Scale) at Screening
7. Patient who has WOMAC score ≥ 1000 at Screening
8. No improvement with persisting knee pain at least for 12 weeks (3 months) by nonoperational therapy before Screening

Exclusion Criteria:

1. Patients who have pregnancy plans within this trial period or childbearing age patients who do not agree to maintain contraception status through appropriate contraception methods

   * Appropriate contraception method: Use of condom, contraceptive sponges, foam, diaphragm, intrauterine device etc.
   * Periodic abstinence(e.g. methods of predicting ovulation) and moderation are not considered as appropriate contraception method.
   * Not allowed to use hormonal contraceptives
   * Childbearing age female patients, exclude menopausal female (amenorrhea for more than 24 months after the last menstruation) or female who has no possibility of pregnency by surgical sterilization operation, can participate in this study only determined negative in pregnancy test
2. Pregnant women or lactating mothers
3. Patients with Body Mass Index (BMI) > 35
4. Patients with positive human immunodeficiency (HIV), hepatitis B (HBV), hepatitis C (HCV), syphilis at screening indicative of current of pass infection
5. Patients with other disease including

   * Septic arthritis, Rheumatoid or Inflammatory joint disease, Gout, Reccurent pseudogout, Paget disease, Articular fractures, Ochronosis, Acromegaly, Hemochromatosis, Wilson's disease,Osteochondromatosis, Hereditary disorder, Genetic disorder of collagen
6. Patients who are diagnosed with malignant tumor in the past or present
7. Patients who have clinically significant diseases including

   * Cardiac disorder (Myocardial infarction, Coronary artery bypass graft, Arrhythmia and other severe Cardiac disorder etc.)
   * Resistant hypertension (systolic blood pressure > 160mmHg or diastolic pressure > 100mmHg at Screening)
   * Kidney disease (Chronic renal failure, Glomerulonephritis etc.)
   * Liver disease (Hepatocirrhosis, Fatty liver, acute or chronic liver disease etc.)
   * Endocrinopathy (Thyroiditis, Diabetes insipidus, Cushing disease etc.)
8. Patients who have significant lab abnormalities
9. Patients who have severe pain in other areas that can affect the judgement of knee joint symptom
10. Patients who underwent any arthroscopic surgery on the injection site within 6 months of the screening visit date, or scheduled to perform any surgery during the clinical trial period
11. Patients who received any drug by intra-articular injection(hyaluronic acid or steroid etc.) for treatment within 6 months prior to Screening
12. Patients who experienced as stem cell therapy or blood product injection(PRP, Prolo injection etc.)
13. Patients who received treatment within 14 days prior to Screening including(But, patients who had wash-out-period can participate in this study)

    * Take medicines including composition of Glucosamine, Chondretin sulphate and Diacerhein etc.
    * Take phytotherapeutic agent or Chinese medicine for osteoarthritis
    * Take antiinflammatory analgesic drug, NSAIDs (prescription/nonprescription pharmaceuticals) etc. (Patients who have 3 days of wash-out-period after they took acetaminophen can participate in the study)
    * Take oral steroids
    * Physical therapy or Chinese medical treatment(cupping, acupuncture, moxibustion etc.)
14. Patients with penicillin hypersensitivity reactions
15. Patients with skin diseases or infections in the area of the injection site
16. Patients who have abnormal flail over grade 2 flail knee test of anterior to posterior and varus/valgus lesion at physical examination
17. Patients who have difficulty in taking MRI because of metal materials (cardiac pacemaker or clip of cerebral artery etc.) in their body or claustrophobia -but, patients with metal materials that are not affected by magnetic field can participate in this study
18. Patients who have difficulty in liposuction or local anesthesia
19. Patients who have alcohol, drug abuse history
20. Patients who have severe neurologic and psychiatric disorders that affect clinical trials
21. Patients who had participated in other clinical trials within 12 weeks prior to this study
22. Patients who the principal investigator considers inappropriate for the clinical trial due to any other reasons than those listed above

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Change of Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC) scores from baseline | 12 weeks, 24 weeks
  Pain, stiffness, and physical function of the knee will be measured by the WOMAC score
  * Score range is
    1. 0-20 for Pain
    2. 0-8 for Stiffness
    3. 0-68 for Pysical Function
  * Higher scores on the WOMAC indicate wors pain, stiffness, and functional limitations
Change of Visual Analog Scale (VAS) scores from baseline | 12 weeks, 24 weeks
  Pain of knee will be measured by the 100mm VAS
  -Score range is from 0-4mm(no pain) to 75-100mm(severe pain)

SECONDARY OUTCOMES:
WOMAC 3 subscale score | 12 weeks, 24 weeks
  Pain, stiffness, and physical function of the knee will be measured by the Western Ontario and McMaster Universities (WOMAC)
VAS score | 12 weeks, 24 weeks
  Pain of knee will be measured by the 100mm Visual Analog Scale (VAS)
KOOS | 12 weeks, 24 weeks
  Symptoms, pain and functionality of the knee joint will be evaluated via the Knee Injury and Osteoarthritis Outcome Score (KOOS)
  -Score range is from 0(extreme symptoms) to 100(no symptoms)
SF-36 | 12 weeks, 24 weeks
  The SF(Short Form)-36 Health Survey is a 36-item, patient-reported survey of patient health.
IKDC | 12weeks, 24 weeks
  Symptoms, sports activities, and function of the knee will be measured by the International Knee Documentation Committee (IKDC)
Measuring of Kellgren-Lawrence grade | 12 weeks, 24 weeks
  Measuring of Kellgren-Lawrence grade through X-ray
Measuring of Femoro-tibial anatomical angle(FTA) | 12 weeks, 24 weeks
  Measuring of FTA through X-ray
Measuring of Hip-Knee-Ankle angle(HKA) | 12 weeks, 24 weeks
  Measureing of HKA through X-ray
Measuring of Joint Space Width | 12 weeks, 24 weeks
  measuring Joint Space Width through X-ray
MRI scan | 12 weeks, 24 weeks
  MRI perform to measure Modified WORMS (Whole-Organ Magnetic Resonance Imaging Score)
Use of rescue medication | 12 weeks, 24 weeks
  Frequency and total amount of rescue medication administration will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: KANGIL KIM, M.D., Ph.D., Principal Investigator — KyungHee University Gangdong Hospital; WOOSUK LEE, M.D., Ph.D., Principal Investigator — Gangnam Severance Hospital; SUNCHUL HWANG, M.D., Ph.D., Principal Investigator — Gyeongsang National University Hospital; SANGJUN SONG, M.D., Ph.D., Principal Investigator — Kyunghee University Medical Center; KICHEOR BAE, M.D., Ph.D., Principal Investigator — Keimyung University Dongsan Medical Center; YOUNGWAN MOON, M.D., Ph.D., Principal Investigator — Samsung Medical Center; JUHONG LEE, M.D., Ph.D., Principal Investigator — Chonbuk National University Hospital; HANJUN LEE, M.D., Ph.D., Principal Investigator — Chunang University Hospital; EUISUNG CHOI, M.D., Ph.D., Principal Investigator — Chungbuk National University Hospital; YONG IN, M.D., Ph.D., Principal Investigator — Seoul St. Mary's Hospital; KWANKYU PARK, M.D., Ph.D., Principal Investigator — Yonsei University; OOGJIN SHON, M.D., Ph.D., Principal Investigator — Yeungnam University Hospital; MYUNGCHUL LEE, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (13):
- South Korea (13):
  - Chungbuk National University Hospital, Cheongju-si
  - Yeungnam University Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Chonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Kyunghee University Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Seoul
  - KyungHee University Gangdong Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Chunang University Hospital, Seoul

REFERENCES:
- [Derived] Kim KI, Lee MC, Lee JH, Moon YW, Lee WS, Lee HJ, Hwang SC, In Y, Shon OJ, Bae KC, Song SJ, Park KK, Kim JH. Clinical Efficacy and Safety of the Intra-articular Injection of Autologous Adipose-Derived Mesenchymal Stem Cells for Knee Osteoarthritis: A Phase III, Randomized, Double-Blind, Placebo-Controlled Trial. Am J Sports Med. 2023 Jul;51(9):2243-2253. doi: 10.1177/03635465231179223. Epub 2023 Jun 21. PMID 37345256